CLINICAL TRIAL: NCT02110797
Title: Osteoporosis in RETT Syndrome. Understanding the Mechanisms and Identification of Biomarkers.
Brief Title: Osteoporosis in RETT Syndrome
Acronym: OSRETT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P071230
Record Dates: First submitted 2014-04-02; First posted 2014-04-10 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: RETT Syndrome With Proven MECP2 Mutation
Keywords: RETT syndrome; MECP2; Osteoporosis; RANK-ligand; osteoprotegerin
MeSH Terms: conditions — Rett Syndrome; Osteoporosis | interventions — Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RETT patients (Other)
  Interventions: Other: biological markers and evaluation of the mineral density at the lumber spine using DEXA

INTERVENTIONS:
Other: biological markers and evaluation of the mineral density at the lumber spine using DEXA

SUMMARY:
Based on our clinical observations, many girls with RETT syndrome, a severe neuro-developmental encephalopathy, suffer from osteoporosis which can appear at a very early age (before age 10) and can lead to fractures, pain and a limitation in mobility. Few epidemiological studies have estimated the frequency of osteoporosis in girls with RETT syndrome and showed that they are more exposed then children with other neuro-developmental diseases with a same degree of neurological handicap. However, the mechanisms that lead to early osteoporosis in RETT syndrome remain unknown. Mutations in the MECP2 gene are found in 95% of RETT patients and preliminary experimental studies have shown that this can lead to abnormal expression of the gene that codes for osteoprotegerin, a protein implicated in bone remodelling by interacting with RANK-ligand.

In order to identify risk factors of osteoporosis in RETT syndrome and to understand the pathophysiological mechanisms the study protocol includes:

1. Clinical evaluation of bone health (history of bone fractures, pain, nutritional status, pubertal stage, daily caloric/calcium intake, anti-epileptic drugs, walking ability, vitamin D satus)
2. evaluation of the mineral density at the lumber spine using DEXA
3. measuring concentrations of osteoprotegerin and RANK-ligand

DETAILED DESCRIPTION:
Based on our clinical observations, many girls with RETT syndrome, a severe neuro-developmental encephalopathy, suffer from osteoporosis which can appear at a very early age (before age 10) and can lead to fractures, pain and a limitation in mobility. Few epidemiological studies have estimated the frequency of osteoporosis in girls with RETT syndrome and showed that they are more exposed to osteoporosis then children with other neuro-developmental diseases with a same degree of neurological handicap. However, the mechanisms that lead to early osteoporosis in RETT syndrome remain unknown.

Mutations in the MECP2 gene are found in 95% of RETT patients. Preliminary experimental studies on the transcriptional consequences of MECP2 mutations showed that the expression of 13 genes were significantly dysregulated and one of them is the gene that codes for osteoprotegerin, a soluble receptor that binds to RANK-ligand. RANK-ligand is an osteoclastic differentiation factor expressed by osteoblasts.

In order to identify risk factors of osteoporosis in RETT syndrome and to understand the pathophysiological mechanisms the study protocol includes:

1. Clinical evaluation of bone health (history of bone fractures, pain, nutritional status, pubertal stage, daily caloric/calcium intake, anti-epileptic drugs, walking ability, vitamin D status)
2. evaluation of the mineral density at the lumber spine using DEXA
3. measuring concentrations of osteoprotegerin and RANK-ligand

ELIGIBILITY:
Inclusion Criteria:

* RETT syndrome
* MECP2 mutation

Exclusion Criteria:

* no identified MECP2 mutation
* history of drugs that interfere with bone metabolism

Ages: 5 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2009-12-10 (Actual); Primary Completion 2014-06-06 (Actual); Study Completion 2014-06-06 (Actual)

PRIMARY OUTCOMES:
osteoporosis in RETT patients | Day 0
  Correlation between clinical/biological risk factors and mineral density and osteoporosis in RETT patients

SECONDARY OUTCOMES:
Biological Mechanisms of osteoporosis | Day 0
  RANK-ligand and osteoprotegerin concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Linglart, MD, PhD, Principal Investigator — Kremlin Bicêtre hospital
Locations (1):
- Kremlin bicêtre, Bicêtre, France